CLINICAL TRIAL: NCT02974413
Title: Effectiveness of Self-care Rests on Knowledge, Self-care and Cardiometabolic Control of Adult Men With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Maringá (Other)
Responsible Party: Principal Investigator, Guilherme Oliveira de Arruda, PhD Student, Universidade Estadual de Maringá
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: State University of Maringá
Record Dates: First submitted 2016-08-08; First posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

ARMS (2):
- Intervention (Experimental): The intervention to be performed will be based on the principles and steps of supported self-care, guided by Behavior Change Protocol (Behavior Change Protocol - BCP) and consists of an educational program with quarterly meetings, and individual at home, through home visits, and group in the Basic Health Unit (BHU), in addition to telephone monitoring in the interval between two meetings. This intervention will be applied together adult men with type 2 diabetes who are randomized in the intervention group (IG) for six months. Thus, these men will take part in three meetings, individual or group, and will receive four telephone calls in between the face meetings. Our objective is to draw with this intervention by the participant, an individual plan of self-care, based on concretras goals and supports you in the implementation of this plan, in order to improve their self-efficacy in self-care and therefore glycemic control.
  Interventions: Behavioral: self-care supported
- Control (No Intervention): The study will also include a Control Group (CG), and the participants of this group will participate in conversation circles at the beginning and the end of the six month follow-up.

INTERVENTIONS:
Behavioral: self-care supported — The intervention to be performed will be based on the principles and steps of supported self-care, guided by Behavior Change Protocol (Behavior Change Protocol - BCP) and consists of an educational program with quarterly meetings, and individual at home, through home visits, and group in the Basic Health Unit (BHU), in addition to telephone monitoring in the interval between two meetings. This intervention will be applied together adult men with type 2 diabetes who are randomized in the intervention group (IG) for six months. Thus, these men will take part in three meetings, individual or group, and will receive four telephone calls in between the face meetings. Our objective is to draw with this intervention by the participant, an individual plan of self-care, based on concretras goals and supports you in the implementation of this plan, in order to improve their self-efficacy in self-care and therefore glycemic control.The study will also include a Control Group (CG).
  Arms: Intervention

SUMMARY:
This research project has the main objective to analyze the benefits of self-care supported for adult men with Diabetes Mellitus. Treat yourself will randomized-controlled clinical study, randomized cluster to be developed with men aged between 40 and 70 years who have type 2 diabetes and are registered with the Health Strategy teams of the Municipality of Family Maringa. The recruited subjects will be randomly allocated into two groups: intervention group and control group. In the first, individuals will participate in a self-care intervention supported by a nurse, based on supported self-care and behavior change protocol; and second, individuals participate in conversation circles and will have the assistance normally provided by health services. The follow-up will take place for six months and will be collected information: socioeconomic, demographic, behavioral health, complications, laboratory and anthropometric. It is intended, through this study, demonstrate the effectiveness of this type of intervention, user-centric, on the health of men with DM, reinforcing this option of choice for professionals and users within the Primary Health Care (PHC).

ELIGIBILITY:
Inclusion Criteria:

* Having medical diagnosis of DM2;
* Being male;
* Age between 20 and 59 years;
* Is domiciled in the city of Maringa in the FHS coverage area; Being part of the ESF families register.
* Being able to answer the questions of data collection instruments;
* Relate visual ability , hearing and locomotor to perform self-care;
* Have telephone contact (mobile or fixed) for monitoring the program.

Exclusion Criteria:

* Present lesions in target organs (brain, heart, kidneys, eyes) or comorbidities/complications resulting from diabetes, recorded in medical records, such as chronic renal failure;
* Have psychological or other disorders , registered in the medical records, and that compromise the understanding of the study, who do not agree or do not have availability to participate in the intervention;
* Moving to another location that does not have coverage of the ESF, or even to another city.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Baseline and six months
  Change in glycemic control between baseline and six months: should be determined by the values of glycated hemoglobin, which will be compared between the two moments (baseline and six months).

SECONDARY OUTCOMES:
Self-care attitudes | Baseline and six months
  Self-care attitudes: measured from QAD questionnaire ( Self Care Questionnaire in Diabetes). For the analysis of adherence to the questionnaire items, they will be parameterized in number of days per week, from zero to seven, zero being the least desirable and seven to more favorable situation, with the exception of items the size specific power that question assessing the consumption of foods rich in fat and sweets, for which the values are reversed, Ie in relation to these foods, the higher the score, or the number of days, the less desirable it is. It will be evaluated by the average number of days. comparisons will be made between the beginning and at the end of the intervention.
Self-efficacy (or Empowerment) | Baseline and six months
  Self-efficacy (or Empowerment): measured from the self-efficacy scale in diabetes - short version (EAD -VC). The questionnaire addresses the training for the care of diabetes. Eight statements for which the respondent demonstrate their level of agreement, using a Likert scale of five points that part of "strongly disagree" (one point ) to" strongly agree" (five points). The overall score is calculated by the average of the scores of each of the eight items. It is considered high a score of 3.8-5.0, an average of 2.4-3.7 and low at 1-2.3. comparisons will be made between the beginning and at the end of the intervention.
Psychological adjustment | Baseline and six months
  Psychological adjustment: We used the ATT -19 instrument, which contains 19 items and describes the emotional responses of the DM. Each statement is answered with the help of a kind of scale Likert five points, from " Strongly disagree" to" Strongly agree". TTA -19 Apontuação will 19-95 points. To achieve a positive attitude about DM, the user needs to achieve a minimum score of 70 points. comparisons will be made between the beginning and at the end of the intervention.
Knowledge about diabetes | Baseline and six months
  Knowledge about diabetes: test was used which has a total score of 15 points, addressing the knowledge of the DM. The DKN-A is associated with psychological, hypoglycemia, insulin, food groups, replacement of food, DM management and general principles of care of the disease. To show a satisfactory knowledge of the DM, the user needs to do at least 8 points. comparisons will be made between the beginning and at the end of the intervention.
Clinical indicators of cardiometabolic control | Baseline and six months
  Clinical indicators of cardiometabolic control (Blood Pressure, Body Fat Percentage, CA, WHR, BMI, weight, fasting glucose, triglycerides, total cholesterol, HDL, LDL, Creatinine Plasma). comparisons will be made between the beginning and at the end of the intervention.
Height | Baseline and six months
  Height in meters (m), measured by portable stadiometer.
Weight | Baseline and six months
  Weight in kilograms (kg), measured by means of a portable scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual de Maringá, Maringá, Paraná, Brazil